CLINICAL TRIAL: NCT02155231
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Study on Anal Human Papillomavirus Infection and Anal Intraepithelial Neoplasia Among Men Who Have Sex With Men in Indonesia, Malaysia, and Thailand
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Verein Aids Life through TREAT Asia (Unknown)
Responsible Party: Sponsor
Other Study IDs: Anal HPV and AIN among MSM
Record Dates: First submitted 2014-05-28; First posted 2014-06-04 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HPV Testing
Keywords: Male with history of anal sex with men or previous participants of the MSM VCT study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- previous enrolled
- New Enrolled

SUMMARY:
OBJECTIVES

1. To determine the prevalence and incidence of anal HPV infection, including infection with high-risk HPV types, among MSM in Indonesia, Malaysia, and Thailand.
2. To study the prevalence and incidence of HGAIN among these MSM.
3. To evaluate risk factors, including HIV status, for anal high-risk HPV infection and HGAIN among these MSM.

Study population An approximately 75 HIV-positive and 75 HIV-negative MSM who attended the study clinic in Kuala Lumpur, Jakarta, and Bangkok will be enrolled. The study will also enroll 185 HIV-positive and 95 HIV-negative MSM who are previous participants of the MSM VCT study. There will be approximately 260 HIV-positive and 170 HIV-negative MSM in total in this study.

DETAILED DESCRIPTION:
This is a prospective cohort study that will newly enroll approximately 150 MSM in Kuala Lumpur, Jakarta, and Bangkok and follow them prospectively with a group of 280 MSM who are previous participants of a study entitled "Multidisciplinary services to enhance HIV testing and linkage to care among MSM" (MSM VCT study) in Jakarta, Bali, and Bangkok. Newly enrolled MSM will have three study visits at baseline, month 6, and at month 12. MSM who are previous participants of the MSM VCT study will only have one study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male with history of anal sex with men or previous participants of the MSM VCT study.
2. Age 18 years old or older.
3. Indonesian or Malaysian or Thai citizen as identified by the Indonesian or Malaysian or Thai National Identification card.
4. Willing to provide location or contact information and allow contact.
5. Available for follow-up for the planned study duration.
6. Understand the study and sign informed consent form.

Exclusion Criteria:

1. History of prior treatment for anal cancer OR had anal cytology or high-resolution anoscopy or infrared coagulation within 12 months prior to enrollment OR had trichloroacetic acid or podophyllin application of the intraanal area in the past month OR evidence of active concurrent intraanal or perianal bacterial or herpes simplex infection.
2. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with ability to give informed consent.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An approximately 75 HIV-positive and 75 HIV-negative MSM who attended the study clinic in Kuala Lumpur, Jakarta, and Bangkok will be enrolled. The study will also enroll 185 HIV-positive and 95 HIV-negative MSM who are previous participants of the MSM VCT study. There will be approximately 260 HIV-positive and 170 HIV-negative MSM in total in this study.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
prevalence and incidence of anal HPV infection, including infection with high-risk HPV types, among MSM in Indonesia, Malaysia, and Thailand. | December 1,2014 (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand